CLINICAL TRIAL: NCT03650842
Title: Changes in Cerebral Oxygenation During Laparoscopic Pyloromyotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB16-00199
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Pyloric Stenosis
MeSH Terms: conditions — Pyloric Stenosis | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Laparoscopic pyloromyotomy (Experimental): Infants undergoing laparoscopic pyloromyotomy.
  Interventions: Device: Near infrared spectroscopy (NIRS)

INTERVENTIONS:
Device: Near infrared spectroscopy (NIRS) — One monitor will be placed on the forehead to measure cerebral oxygenation and a second over the lower back to measure tissue (muscle or renal) oxygenation.

SUMMARY:
A prospective study that will assess the effect of laparoscopy on tissue oxygenation in the patients undergoing a laparoscopic pyloromyotomy at Nationwide Children's Hospital. Tissue oxygenation will be assessed non-invasively using near infrared spectroscopy, a device that is commonly used in our operating rooms to assess cerebral and tissue oxygenation.

DETAILED DESCRIPTION:
This prospective study will include 50 patients under the age of 18 years who are having laparoscopic pyloromyotomy. There will be no change in the anesthetic or perioperative care of these patients. Tissue and cerebral oxygenation will be monitored using near infrared spectroscopy (NIRS). Prior to anesthetic induction, the NIRS monitor will be placed on the forehead. The device is non-invasive like pulse oximetry using a non-painful adhesive sticker. The device can be applied to different sites on the body to measure cerebral, tissue or even organ oxygenation. For the purpose of the study, the investigators will place one monitor on the forehead to measure tissue oxygenation and a second over the lower back to measure tissue (muscle or renal) oxygenation. These devices are used routinely in the operating room and the cardiothoracic intensive care unit for cardiac patients. Although not used on every surgical procedure, NIRS monitoring can be used on all patients who are undergoing major surgical procedures. Tissue and cerebral oxygenation will be recorded continuously starting just prior to anesthetic induction until the completion of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children at Nationwide Children's Hospital under the age of 18 years who are having laparoscopic pyloromyotomy

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamata M, Hakim M, Walia H, Tumin D, Tobias JD. Changes in cerebral and renal oxygenation during laparoscopic pyloromyotomy. J Clin Monit Comput. 2020 Aug;34(4):699-703. doi: 10.1007/s10877-019-00356-2. Epub 2019 Jul 19. PMID 31325010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laparoscopic Pyloromyotomy
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Laparoscopic Pyloromyotomy: Patients undergoing laparoscopic pyloromyotomy.
Arm/Group | Laparoscopic Pyloromyotomy
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: days] | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25
Weight [Mean (Standard Deviation); unit: kilograms] | 4 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Regional Oxygen Saturation (rSO2)
Description: Near-infrared spectroscopy (NIRS model INVOS 5100; Covidien, Minneapolis, MN, USA) with sensors (Neonate SomaSensor® CNN; Covidien, Minneapolis, MN, USA) placed on the forehead.
Time Frame: At time of incision
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Laparoscopic Pyloromyotomy
Number analyzed (Participants) | 25
percentage of oxygen | 81 (12)

2. Primary Outcome: Cerebral Regional Oxygen Saturation (rSO2)
Description: as for outcome 1
Time Frame: At the end of laparoscopy
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Laparoscopic Pyloromyotomy
Number analyzed (Participants) | 25
percentage of oxygen | 76 (16)

3. Primary Outcome: Renal Regional Oxygen Saturation (rSO2)
Description: Near-infrared spectroscopy (NIRS model INVOS 5100; Covidien, Minneapolis, MN, USA) with sensors (Neonate SomaSensor® CNN; Covidien, Minneapolis, MN, USA) placed on the left posterior-lateral flank.
Time Frame: At time of incision
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Laparoscopic Pyloromyotomy
Number analyzed (Participants) | 25
percentage of oxygen | 83 (11)

4. Primary Outcome: Renal Regional Oxygen Saturation (rSO2)
Description: as for outcome 3
Time Frame: At the end of laparoscopy
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Laparoscopic Pyloromyotomy
Number analyzed (Participants) | 25
percentage of oxygen | 77 (20)

ADVERSE EVENTS:
Time Frame: Adverse events collected on day of surgery only.
Arm/Group | Laparoscopic Pyloromyotomy
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT03650842/Prot_SAP_000.pdf